CLINICAL TRIAL: NCT03198481
Title: Protocol for Patient-Centered Versus Physician-Centered Counseling Video for Midurethral Slings an RCT
Brief Title: Patient-Centered Versus Physician-Centered Counseling MidUrethral Sling Videos
Acronym: MUVi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-058
Record Dates: First submitted 2017-05-25; First posted 2017-06-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Stress Urinary Incontinence; Satisfaction
Keywords: midurethral sling; movie; preparedness; Video Counseling
MeSH Terms: conditions — Urinary Incontinence, Stress; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-Centered Counseling Video Group (Active Comparator): MUS video utilizing a patient mentor.
  Interventions: Behavioral: Patient-Centered Counseling Video
- Physician Counseling Video Group (Active Comparator): MUS video by a physician.
  Interventions: Behavioral: Physician Counseling Video

INTERVENTIONS:
Behavioral: Patient-Centered Counseling Video — Patients will watch a patient-centered education video regarding MUS prior to standard pre-operative counseling.
  Arms: Patient-Centered Counseling Video Group
Behavioral: Physician Counseling Video — Patients will watch a physician-centered video regarding MUS prior to standard pre-operative counseling.
  Arms: Physician Counseling Video Group

SUMMARY:
The decision making process for stress incontinence surgery is complex. A key gap in the literature is how to improve patient preparedness and satisfaction for mid-urethral sling (MUS) surgery that is reproducible and low cost. Multimedia can assist in bridging this gap. The specific aims of the proposed research: (1) is to develop two videos to counsel patients who have elected to undergo a MUS surgery. One video will be created from a patient-centered perspective using peers as counselors. The second will employ a traditional counseling approach; (2) To compare the impact of multimedia counseling between women randomized to a patient-centered counseling versus a traditional counseling video. The investigators will recruit patients who present with stress urinary incontinence who elect to undergo a MUS procedure. Women will be randomized during their pre-operative visit to watch the patient-centered or traditional counseling video before they are counseled regarding their upcoming MUS surgery in the usual manner. The investigators anticipate women randomized to a patient centered-video will report higher satisfaction, less decisional regret, greater preparedness, and less anxiety as measured by validated scales. Successful completion will improve understanding of patient's needs and will allow development of improved educational tools readily available to the AUGS community.

DETAILED DESCRIPTION:
Management of Pelvic Floor Disorders (PFDs) is individualized according to a patient's symptomatology and quality of life. Although conservative measures exist, patients may elect for surgical management. The decision making process for surgery is complex. It is well documented that patient's lack understanding prior to their surgical procedures. Preparedness for MUS surgery is related to a patient's comprehension of the purpose, risks, benefits, and complications. Patients who are more prepared prior to surgery have been proven to have greater postoperative satisfaction. Therefore, it is essential to improve patients' preparedness and enhance patients' understanding of realistic expectations of post-operative outcomes.

The investigators long-term goal is to improve patient-centered preparedness and satisfaction when considering surgery. Previous studies by the Preliminary Study of Peer Support Groups and Pelvic Floor Disorders have demonstrated trends in improvement for preparedness and decision conflict with the use of peer focus groups. However, peer support groups are a costly process and there may be many barriers to participation.

A key gap in the literature is how to improve patient preparedness for surgery and improve satisfaction through the use of peer counseling in a manner that is convenient for patients, reproducible and low cost. Technological advances with multimedia may assist in bridging this gap. With ease-of-access to mobile electronic devices, videos are effective tools to prepare patients for surgery. The purpose of this randomized controlled clinical trial is to determine if a patient-centered video improves satisfaction and preparedness compared to a physician-centered video.

The first objective of this research is to develop two videos to counsel patients who have elected to undergo a MUS procedure. One video will be created from a physician-centered approach. The second video will be a patient-centered perspective. The second objective of this research is to compare the impact of video counseling between women randomized to a physician-centered versus a patient-centered video. The central hypothesis is that women randomized to a patient-centered video will report higher scores of satisfaction and preparedness than women randomized to the physician-centered video.

Specifically, our aims for this study are:

1. To create two videos to be used to counsel patients who have elected to undergo a MUS procedure. One video will present the risks, benefits and alternatives to MUS surgery by a physician, mimicking traditional counseling prior to surgery. The second video will explain the risks, benefits and alternatives to the MUS surgery utilizing a patient mentor who has undergone the MUS procedure and will describe the patients' perception of the information. The patient-centered video will also include topics that have previously been identified by focus groups as important patient-centered aspects of pre-surgical counseling.
2. To compare the impact of video counseling between women randomized to a physician-centered video and a patient-centered video. Hypothesis: Women randomized to a patient centered-video will report higher satisfaction and preparedness as measured by validated scales. They will have higher scores on the Post-operative preparedness questionnaire (PPQ), Preparedness Scale and the Surgical Decision Satisfaction (SDS-PFD) questionnaire; and lower scores on the Decision Regret Scale (DRS-PFD) questionnaire than women randomized to view the physician-centered video prior to undergoing mid-urethral sling surgery.
3. To compare a women's decisional conflict post-operatively in women randomized to the physician-centered video and the patient-centered video. Hypothesis: There is a reduction of decisional conflict in women randomized to the patient-centered video.
4. To determine if there are differences in anxiety scores in women who watch the patient-centered video versus the physician centered video. Hypothesis: Anxiety scores measured by the State Trait Anxiety Inventory (STAI: Y-6 Item) questionnaire are decreased by a pre-operative patient-centered counseling video.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are ≥ 18 years of age
2. Planning to undergo a midurethral sling procedure
3. Either stress urinary incontinence (SUI) or mixed urinary incontinence (MUI) with a positive cough stress test or SUI documented on urodynamic testing
4. English speaking

Exclusion Criteria:

1. Those who desire a concomitant POP Surgery
2. Inability to speak/understand English
3. Prior midurethral sling performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Patient preparedness | Change from baseline at the 6 weeks post-operative visit
  The objective is to compare patient preparedness between women in the patient-centered and physician centered video group. The investigators hypothesize that subjects in the patient-centered video group will report higher preparedness pre-operative and 6 weeks post-operative on the Patient Preparedness Questionnaire (PPQ). The investigators will assess the level of pre-operative and post-operative preparedness according to each preparedness question on the Patient Preparedness Questionnaire (PPQ).

SECONDARY OUTCOMES:
Patient Satisfaction | Change from baseline at the 6 weeks post-operative visit
  The objective is to compare patient satisfaction between women in the patient-centered and physician centered video group. The investigators hypothesize that subjects in the patient-centered video group will report higher satisfaction scores pre-operative and 6 weeks post-operative. Satisfaction will be measured by the Satisfaction with Decision Scale-Pelvic Floor Disorders (SDS-PFD) at her pre-operative visit and at the subjects 6 week visit.
Decision Regret | 6 weeks post-operative visit
  The objective is to compare patient decision regret between women in the patient-centered and physician centered video group. The investigators hypothesize that subjects in the patient-centered video group will report less decision regret at their 6 weeks post-operative visit. Decision regret will be evaluated using the Decision Regret Scale-Pelvic Floor Disorders (DRS-PFD) and at the subjects 6 week visit.

OTHER OUTCOMES:
Patient Decisional Conflict | Baseline
  To compare a women's decisional conflict pre-operatively in women randomized to the patient-centered and physician centered video using the Decisional Conflict Score (DCS) Questionnaire.
Patient Anxiety | Change from baseline at the 6 weeks post-operative visit
  To determine if there are differences in anxiety scores in women who watch the patient-centered video versus the physician centered video using the STAI: Y-6 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yuko M Komesu, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - Dell Medical School at University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reading AE. Psychological preparation for surgery: patient recall of information. J Psychosom Res. 1981;25(1):57-62. doi: 10.1016/0022-3999(81)90084-2. No abstract available. PMID 7277269
- [Background] Pool JJ. Expected and actual knowledge of hospital patients. Patient Couns Health Educ. 1980 3d Quart;2(3):111-7. doi: 10.1016/s0738-3991(80)80051-6. No abstract available. PMID 10249187
- [Background] Kenton K, Pham T, Mueller E, Brubaker L. Patient preparedness: an important predictor of surgical outcome. Am J Obstet Gynecol. 2007 Dec;197(6):654.e1-6. doi: 10.1016/j.ajog.2007.08.059. PMID 18060968
- [Background] Brubaker L, Litman HJ, Rickey L, Dyer KY, Markland AD, Sirls L, Norton P, Casiano E, Paraiso MF, Ghetti C, Rahn DD, Kusek JW. Surgical preparation: are patients "ready" for stress urinary incontinence surgery? Int Urogynecol J. 2014 Jan;25(1):41-6. doi: 10.1007/s00192-013-2184-x. Epub 2013 Aug 3. PMID 23912506
- [Background] Mancuso CA, Salvati EA, Johanson NA, Peterson MG, Charlson ME. Patients' expectations and satisfaction with total hip arthroplasty. J Arthroplasty. 1997 Jun;12(4):387-96. doi: 10.1016/s0883-5403(97)90194-7. PMID 9195314
- [Background] Firoozi F, Gill B, Ingber MS, Moore CK, Rackley RR, Goldman HB, Vasavada SP. Increasing patient preparedness for sacral neuromodulation improves patient reported outcomes despite leaving objective measures of success unchanged. J Urol. 2013 Aug;190(2):594-7. doi: 10.1016/j.juro.2013.03.025. Epub 2013 Mar 14. PMID 23499745
- [Background] Fultz NH, Burgio K, Diokno AC, Kinchen KS, Obenchain R, Bump RC. Burden of stress urinary incontinence for community-dwelling women. Am J Obstet Gynecol. 2003 Nov;189(5):1275-82. doi: 10.1067/s0002-9378(03)00598-2. PMID 14634553
- [Background] Paraiso MF, Muir TW, Sokol AI. Are midurethral slings the gold standard surgical treatment for primary genuine stress incontinence? J Am Assoc Gynecol Laparosc. 2002 Nov;9(4):405-7. doi: 10.1016/s1074-3804(05)60510-5. No abstract available. PMID 12386347
- [Background] McFadden BL, Constantine ML, Hammil SL, Tarr ME, Abed HT, Kenton KS, Sung VW, Rogers RG. Patient recall 6 weeks after surgical consent for midurethral sling using mesh. Int Urogynecol J. 2013 Dec;24(12):2099-104. doi: 10.1007/s00192-013-2136-5. Epub 2013 Jul 2. PMID 23818127
- [Background] Dmochowski RR, Blaivas JM, Gormley EA, Juma S, Karram MM, Lightner DJ, Luber KM, Rovner ES, Staskin DR, Winters JC, Appell RA; Female Stress Urinary Incontinence Update Panel of the American Urological Association Education and Research, Inc; Whetter LE. Update of AUA guideline on the surgical management of female stress urinary incontinence. J Urol. 2010 May;183(5):1906-14. doi: 10.1016/j.juro.2010.02.2369. Epub 2010 Mar 29. PMID 20303102
- [Background] Ellett L, Villegas R, Beischer A, Ong N, Maher P. Use of a multimedia module to aid the informed consent process in patients undergoing gynecologic laparoscopy for pelvic pain: randomized controlled trial. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):602-11. doi: 10.1016/j.jmig.2014.01.002. Epub 2014 Jan 23. PMID 24462856
- [Background] Dawdy K, Bonin K, Russell S, Ryzynski A, Harth T, Townsend C, Liu S, Chu W, Cheung P, Chung H, Morton G, Vesprini D, Loblaw A, Cao X, Szumacher E. Developing and Evaluating Multimedia Patient Education Tools to Better Prepare Prostate-Cancer Patients for Radiotherapy Treatment (Randomized Study). J Cancer Educ. 2018 Jun;33(3):551-556. doi: 10.1007/s13187-016-1091-5. PMID 27526692

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03198481/Prot_SAP_000.pdf